CLINICAL TRIAL: NCT04732598
Title: A Phase III, Randomized Study of Bevacizumab and Paclitaxel in Combination with Atezolizumab As a Treatment for Patients with Locally Advanced Unresectable or Metastatic Hormone Receptor-positive HER2 Negative Breast Cancer
Brief Title: A Phase III Study of Bevacizumab and Paclitaxel in Combination with Atezolizumab As a Treatment for Locally Advanced Unresectable or Metastatic Hormone Receptor-positive HER2 Negative Breast Cancer
Acronym: AMBITION
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Japanese Foundation for Cancer Research (Other)
Collaborators: Chugai Pharmaceutical (Industry)
Responsible Party: Principal Investigator, Fumikata Hara, M.D., Ph.D. Chief, Breast Medical Oncology, Aichi Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JCOG1919E
Record Dates: First submitted 2021-01-28; First posted 2021-02-01 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Paclitaxel; Bevacizumab; atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (Active Comparator)
  Interventions: Drug: Paclitaxel + bevacizumab therapy
- Arm B (Experimental)
  Interventions: Drug: Paclitaxel + bevacizumab + atezolizumab

INTERVENTIONS:
Drug: Paclitaxel + bevacizumab therapy — The following regimen will be continued as a 28-day course until disease progression or the criteria for treatment discontinuation are met.
  [Paclitaxel] 90mg/m^2, day1,8,15, IV [Bevacizumab] 10mg/kg, day1,15, IV
  Arms: Arm A
Drug: Paclitaxel + bevacizumab + atezolizumab — The following regimen will be continued as a 28-day course until disease progression or the criteria for treatment discontinuation are met.
  [Atezolizumab] 840 mg/body, day 1,15, IV [Paclitaxel] 90mg/m^2, day1,8,15, IV [Bevacizumab] 10mg/kg, day1,15, IV
  Arms: Arm B

SUMMARY:
JCOG1919E (AMBITION) is a randomized, open-label, phase 3 trial to evaluate efficacy and safety of bevacizumab and paclitaxel in combination with atezolizumab comparing to bevacizumab and paclitaxel in patients with HR-positive HER2 negative metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically diagnosed as breast cancer (invasive cancer).
2. Histologically diagnosed as hormone receptor positive (at least one of ER and PgR is positive) and HER2 negative. However, if there are multiple specimens, the histological results of the most recent specimen that meets the eligibility criteria 1. and 2. should be used.
3. Diagnosed with advanced recurrent breast cancer (either unresectable locally advanced breast cancer, recurrent breast cancer, or Stage IV breast cancer).
4. Age 20 years or older on the date of registration. Either male or female are acceptable.
5. ECOG performance status (PS) of 0-2.
6. Patients must have measurable lesions.
7. Hormone refractory[*a] or life-threatening metastases [*b].

   1. Hormone refractory: Recurrence within 2 years after the start of postoperative endocrine therapy, or progression within 6 months of endocrine therapy for advanced recurrent breast cancer.
   2. Life-threatening metastases: Symptomatic metastases that require symptomatic relief through urgent tumor shrinkage. Examples include multiple liver metastases, lung metastases, carcinomatous pleurisy, and carcinomatous lymphangitis.
8. PD-L1 status has been confirmed by a central measurement institute.
9. No active brain metastases that require treatment.
10. No history of prior chemotherapy treatment for advanced or recurrent breast cancer. However, in case that a history of preoperative/postoperative chemotherapy including paclitaxel or docetaxel, it is acceptable if at least 6 months have passed since the last dose.
11. The most recent laboratory test within 14 days prior to enrollment (the same day of the week two weeks prior to the date of enrollment is acceptable) must meet all of the following

    1. Neutrophil count ≥1,500/mm^3
    2. Hemoglobin ≥ 9.0 g/dL (No blood transfusion within 14 days prior to the date of blood collection for the test used for registration)
    3. Platelet count ≥10×104/mm^3
    4. Total bilirubin ≤ 1.5 mg/dL
    5. AST ≤ 100 IU/L (≤ 150 IU/L if liver metastasis is present)
    6. ALT ≤ 100 IU/L (≤ 150 IU/L in case of liver metastasis)
    7. Serum creatinine ≤1.2 mg/dL
    8. PT-INR ≤ 1.5, but PT-INR ≤ 3.0 if the patient is taking anticoagulants such as warfarin prophylactically.
    9. Urine protein (test paper method) of 1+ or less
12. For women of childbearing potential [*a], consent for contraception from the time of obtaining consent until at least 6 months after completion of the protocol treatment. For lactating patients, the patient agrees not to breastfeed from the start of protocol treatment until at least 6 months after the end of protocol treatment. For men, they agree to use contraception from the start of protocol treatment until at least 6 months after the end of protocol treatment [*b].

    1. Women of childbearing potential: Women who have experienced menarche, have not undergone sterilization (hysterectomy or bilateral oophorectomy), and have not undergone menopause. Menopause is defined as the absence of menstruation for more than 12 months without another medical reason such as drug administration.
    2. Examples of contraceptive methods: condoms, pessaries, oral contraceptives, use of intrauterine devices, etc.
13. The patient's written consent to participate in the study has been obtained.

Exclusion Criteria:

1. Active multiple cancer. However, the following are excluded: ①Completely resected cancers: basal cell carcinoma, Stage I spinous cell carcinoma, intraepithelial carcinoma, intramucosal carcinoma, superficial bladder cancer, ② gastrointestinal tract cancer that has been curatively resected by ESD or EMR, and ③ other cancers that have not recurred for more than 5 years.
2. Infectious diseases that require systemic treatment.
3. Complicated active gastrointestinal ulcer.
4. Patients must have poorly controlled hypertension (systolic blood pressure ≥150 mmHg and/or diastolic blood pressure ≥100 mmHg) despite the use of two or more antihypertensive agents.
5. Patients must have symptomatic congestive heart failure, unstable angina, or arrhythmia requiring treatment at the time of enrollment.
6. History of myocardial infarction within 1 year prior to enrollment.
7. Major surgery or incisional biopsy or significant trauma within 28 days prior to enrollment; placement of a CV port is not considered major surgery.
8. Patients with deep vein thrombosis or pulmonary embolism at the time of enrollment, or a history of such within 1 year prior to enrollment.
9. Use of anticoagulants (except aspirin of 324 mg/day or less) within 10 days prior to enrollment.
10. Patients with a history of idiopathic pulmonary fibrosis, organizing pneumonia (bronchiolitis obliterans, etc.), drug-induced pneumonitis, or idiopathic pneumonitis. However, patients with a history of drug-induced pneumonitis who are asymptomatic at the time of enrollment can be enrolled if they undergo regular chest X-ray examinations and careful follow-up including auscultation and medical examination.
11. Findings of active pneumocystitis on chest CT. However, a history of localized radiation pneumonitis (fibrosis) in the irradiation field is inclusible.
12. Patients have been treated with investigational atezolizumab, or other immune checkpoint inhibitors (e.g., anti-PD-1, anti-PD-L1, anti-CTLA-4 antibody drugs), or immunostimulants (e.g., interferon, interleukin-2).
13. Active autoimmune disease, immunodeficiency, or history thereof (e.g., myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener's granulomatosis, Sjogren's syndrome, Guillain-Barré syndrome, multiple sclerosis, etc.). However, the following are inclusible. Patients with autoimmune hypothyroidism who are using a stable dose of thyroid hormone preparations. Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo vulgaris whose symptoms are limited to the skin, and whose rash accounts for less than 10% of the body surface area and is well controlled by topical application of low potency corticosteroids alone. No acute exacerbation of the underlying disease requiring solaren long-wavelength ultraviolet therapy, methotrexate, retinoids, biologics, oral calcineurin inhibitors, high potency or oral corticosteroids within the past 12 months.
14. Patients who have received a live attenuated vaccine within 4 weeks prior to enrollment or are expected to require a live attenuated vaccine within 5 months of completion of protocol treatment.
15. Patients have not recovered from clinically significant toxicity caused by previous therapy, except for alopecia and Grade 1 peripheral neuropathy.
16. Hypersensitivity or contraindication to any component of the therapeutic agent, including macrogol glycerol ricinoleate (Cremophor®), an additive to paclitaxel.
17. Positive for HIV antibodies, HBs antigen, or HCV antibodies (however, if HCV antibodies are positive but HCV-RNA is not detected, it is not excluded).
18. Negative for HBs antigen, positive for HBs antibody or HBc antibody, and positive for HBV-DNA quantification.
19. Women who are pregnant, lactating, or may be pregnant.
20. Patients with psychosis or psychiatric symptoms that interfere with daily life and are judged to be difficult to participate in the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2021-01-21 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (investigator-assessed) | Up to 2years after last patient enrolled

SECONDARY OUTCOMES:
Progression-free survival (blinded independent central review) | Up to 2years after last patient enrolled
Overall survival | Up to 2years after last patient enrolled
Response rate (investigator-assessed) | Up to 2years after last patient enrolled
Duration of response (investigator-assessed) | Up to 2years after last patient enrolled
Response rate (blinded independent central review) | Up to 2years after last patient enrolled
Duration of response (blinded independent central review) | Up to 2years after last patient enrolled
Incidence of adverse events | Up to 2years after last patient enrolled
Incidence of serious adverse events | Up to 2years after last patient enrolled
Incidence of immune-related adverse events | Up to 2years after last patient enrolled
Progression-free survival in PD-L1 positive subpopulation (investigator-assessed) | Up to 2years after last patient enrolled
PD- L1-positive subpopulation | Up to 2years after last patient enrolled
Progression-free survival in the PD-L1-positive subpopulation (investigator-assessed) | Up to 2years after last patient enrolled
Overall survival in the PD-L1-positive subpopulation | Up to 2years after last patient enrolled
Response rate in the PD-L1-positive subpopulation (investigator-assessed) | Up to 2years after last patient enrolled
Response rate in the PD-L1-positive subpopulation (blinded independent central review) | Up to 2years after last patient enrolled

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Institute Hospital of JFCR, Tokyo, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No